CLINICAL TRIAL: NCT01607879
Title: Use of β-hydroxy-β-methylbutyrate to Counteract Loss of Muscle Mass and Strength in Older Men With Prostate Cancer Started on Androgen Deprivation Therapy
Brief Title: Use of β-hydroxy-β-methylbutyrate to Counteract Muscle Loss in Men With Prostate Cancer on Androgen Ablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Kathryn A Bylow, MD, Associate Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00016781
Record Dates: First submitted 2012-04-20; First posted 2012-05-30 (Estimated); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Men; Androgen Deprivation Therapy; Elderly; Geriatric; Nutritional supplementation
MeSH Terms: conditions — Prostatic Neoplasms; Multiple Endocrine Neoplasia Type 1 | interventions — Arginine; Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care ADT + (HMB + AG) (Experimental): Standard of care androgen deprivation therapy plus the nutritional supplement HMB + arginine + glutamine (AG)
  Interventions: Drug: Standard of care ADT + (HMB + arginine + glutamine)
- Standard of care ADT (Active Comparator): Standard of care androgen deprivation therapy
  Interventions: Other: Standard of care ADT

INTERVENTIONS:
Drug: Standard of care ADT + (HMB + arginine + glutamine) — 1 packet of HMB+arginine+glutamine contains 1.5 g of the amino acid metabolite HMB + 7 g arginine and 7 g glutamine.
  Take one packet twice daily for 3 months
  Other Names: Juven
  Arms: Standard of care ADT + (HMB + AG)
Other: Standard of care ADT — Patient will receive standard of care androgen deprivation therapy (ADT) alone
  Other Names: Standard of care androgen deprivation therapy (ADT)
  Arms: Standard of care ADT

SUMMARY:
This is a study of HMB plus amino acids in older men with prostate cancer starting androgen deprivation therapy (ADT). The investigators hypothesize that the use of this nutritional supplementation will decrease the loss of muscle mass and strength that occurs when men start ADT.

DETAILED DESCRIPTION:
It is well established that older patients experience age-related loss of muscle mass and function (sarcopenia), presumably due to an imbalance of protein synthesis versus protein breakdown. In addition, studies have shown that men who start on ADT experience increased muscle protein breakdown and decreased synthesis. β-hydroxy-β-methylbutyrate (HMB), a leucine metabolite, has been shown to slow protein breakdown. When HMB is given with arginine and lysine (which support protein synthesis) in randomized trials, researchers have shown that elderly men and women who receive this nutritional supplementation experience improvement in fat-free mass, strength, functionality and protein synthesis when compared with controls. In addition, patients with advanced cancer who experienced weight loss of at least 5% have also been shown to benefit from HMB, with supplementation resulting in a significant increase of fat-free mass when compared to controls. Thus, it seems reasonable that older men with prostate cancer starting on ADT who experience lean muscle loss as a result of aging and ADT, may achieve some benefit from supplementation with HMB as well. Use of HMB in men with prostate cancer has not been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. Age 60 years or older
3. Patients with asymptomatic or minimally symptomatic prostate cancer for which they are about to start androgen deprivation therapy (ADT) per provider recommendation

   * Asymptomatic or minimally symptomatic (as judged by treating physician) metastases allowed
   * Men receiving ADT for localized prostate cancer are allowed
4. Patient able to give informed consent.

Exclusion Criteria:

1. Patient already on ADT
2. Patients who are visiting clinic for a second opinion only
3. Patients with a diagnosis of dementia
4. Patients with a diagnosis of a neuromuscular disorder (i.e. multiple sclerosis)

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2018-07 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Bylow, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care ADT + (HMB + AG): Standard of care androgen deprivation therapy plus the nutritional supplement HMB + arginine + glutamine (AG)
  Standard of care ADT + (HMB + arginine + glutamine): 1 packet of HMB+arginine+glutamine contains 1.5 g of the amino acid metabolite HMB + 7 g arginine and 7 g glutamine.
  Take one packet twice daily for 3 months
Period: Overall Study
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT
Started | 24 | 24
Completed | 23 | 24
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 10 | 13
  >=65 years | 21 | 14 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (5.6) | 67.4 (5.1) | 69.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 24 | 22 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Composition (Lean Body Mass)
Description: This measure will be the change of lean body mass from baseline reported in kilograms.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT
Number analyzed (Participants) | 24 | 24
Kilogram
  Baseline | 54.93 (8.66) | 57.58 (7.39)
  Change from Baseline | -1.27 (1.42) | -0.60 (2.22)
Statistical Analysis 1: Comparison: Standard of Care ADT + (HMB + AG) vs Standard of Care ADT; Test type: Superiority; p = 0.1497, t-test, 1 sided

2. Secondary Outcome: Change From Baseline of Dorsiflexor Muscle Size in mm^2.
Description: Cross-sectional area of the dorsiflexor muscle will be measured in mm^2 using magnetic resonance imaging. The dorsiflexor muscles at the front of the leg are responsible for lifting the ball of the foot with the heel in contact with the ground. One dorsiflexor muscle in one leg was analyzed per participant.
Time Frame: Baseline and 3 months
Population: Due to unavailability of equipment, only 5 subjects in the HMB+AG group and 8 subjects in the standard ADT therapy group completed both baseline and 3 months follow-up measurements.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT
Number analyzed (Participants) | 5 | 8
mm^2
  Baseline | 1378 (322) | 1348 (177)
  Change at 3 months | -36 (37) | 30 (164)
Statistical Analysis 1: Comparison: Standard of Care ADT + (HMB + AG) vs Standard of Care ADT; Test type: Superiority; p = 0.17, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Strength of the Dorsiflexor Muscle in Kilograms.
Description: Dorsiflexor muscle strength in kilograms will be measured with a custom lower leg ergometer. The dorsiflexor muscles at the front of the leg are responsible for lifting the ball of the foot with the heel in contact with the ground.
Time Frame: Baseline and 3 months
Population: Due to unavailability of equipment, only 5 subjects in the HMB+AG group and 10 subjects in the standard ADT group completed both baseline and 3 month follo-up visits.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT
Number analyzed (Participants) | 5 | 10
kilogram
  Baseline | 17.2 (3.1) | 18.0 (3.0)
  Change at 3 months | -1.0 (5.3) | 1.0 (2.0)
Statistical Analysis 1: Comparison: Standard of Care ADT + (HMB + AG) vs Standard of Care ADT; Test type: Superiority; p = 0.75, t-test, 2 sided

4. Secondary Outcome: Physical Performance Measured Using the Short Physical Performance Battery (SPPB)
Description: The SPPB uses Likert-style ratings for balance, walking speed, and standing test (Guralnik, 2000).
  Balance metric is the ability to hold three standing positions (feet side-by-side; side of the heel of one foot touching the big toe of the other foot; heel of one foot in front of and touching the toes of the other) up to 10 seconds. Inability to hold a position scores '0'. The sum of scores is the Balance Score. Scoring range is 0-4. Higher scores indicate better balance.
  Walking metric is time to walk 8 feet. Faster times score more points. Inability to complete the walk scores '0'. The score range is 0-4. Higher scores indicate better mobility.
  The Standing Test. The subject is asked to stand and sit five times as quickly as possible. Inability to complete five repetitions scores '0'. Shorter times score more points. Scoring range is 0-4. Higher scores indicate better mobility.
  Overall score is the sum of the scores ranging 0 to 12. Higher scores indicate better performance.
Time Frame: Baseline and 3 months
Population: Four subjects in the HMB+AG group and one subject in the standard ADT group did not complete the SPPB test at the 3-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 10.6 (1.6) | 10.7 (1.7)
  3 months: number analyzed (Participants) | 20 | 23
  3 months | 11.1 (1.1) | 11.0 (1.2)
Statistical Analysis 1: Comparison: Standard of Care ADT + (HMB + AG) vs Standard of Care ADT; Test type: Superiority; p = 0.925, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in the Number of Fall Events
Description: This measure will be the change in the number of reported falls from baseline (defined as the 3 months preceding the baseline visit), and the 3 month period beginning after the baseline visit and continuing through 3 months of therapy.
Time Frame: Baseline, 3 months
Population: Three subjects in the HMB+AG group did not report the number of falls at the 3-month follow-up.
Measure: Number; unit: Falls
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT
Number analyzed (Participants) | 24 | 24
Falls
  Baseline | 1 | 0
  Change at 3 months: number analyzed (Participants) | 21 | 24
  Change at 3 months | -1 | 0
Statistical Analysis 1: Comparison: Standard of Care ADT + (HMB + AG) vs Standard of Care ADT; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Standard of Care ADT + (HMB + AG) | Standard of Care ADT
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 2/24
Other Adverse Events (participants affected / at risk) | 8/24 | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care ADT + (HMB + AG) (N=24) | Standard of Care ADT (N=24)
Leukocytes decreased (Investigations) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Transient ischemic attack (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care ADT + (HMB + AG) (N=24) | Standard of Care ADT (N=24)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Face pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hand pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Melanoma
Neoplasm - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic event (Nervous system disorders) | 1 (1) | 0 (0)
Incontinence, Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT01607879/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT01607879/ICF_001.pdf